CLINICAL TRIAL: NCT03105128
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled Induction Study of the Efficacy and Safety of Risankizumab in Subjects With Moderately to Severely Active Crohn's Disease
Brief Title: A Study of the Efficacy and Safety of Risankizumab in Participants With Moderately to Severely Active Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M16-006; 2016-003123-32 (EudraCT Number)
Expanded Access: NCT03914261 (No longer available)
Record Dates: First submitted 2017-04-04; First posted 2017-04-07 (Actual); Results first posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease (CD); Risankizumab; ABBV-066; BI 655066
MeSH Terms: conditions — Crohn Disease | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Risankizumab Dose 1 (Period 1) (Experimental): Participants randomized to receive risankizumab dose 1 administered by intravenous (IV) infusion.
  Interventions: Drug: risankizumab IV
- Risankizumab Dose 2 (Period 1) (Experimental): Participants randomized to receive risankizumab dose 2 administered by intravenous (IV) infusion.
  Interventions: Drug: risankizumab IV
- Placebo (Period 1) (Placebo Comparator): Participants randomized to receive placebo for risankizumab administered by intravenous (IV) infusion.
  Interventions: Drug: placebo for risankizumab
- Risankizumab Dose 1 (Period 2) (Experimental): Participants who received placebo in Period 1 and participants with inadequate response at Week 12 in Period 1 randomized to receive risankizumab dose 1 administered by intravenous (IV) infusion in Period 2.
  Interventions: Drug: risankizumab IV
- Risankizumab Dose 2 (Period 2) (Experimental): Participants with inadequate response at Week 12 in Period 1 randomized to receive risankizumab dose 2 administered by subcutaneous (SC) injection in Period 2.
  Interventions: Drug: risankizumab SC
- Risankizumab Dose 3 (Period 2) (Experimental): Participants with inadequate response at Week 12 in Period 1 randomized to receive risankizumab dose 3 administered by subcutaneous (SC) injection in Period 2.
  Interventions: Drug: risankizumab SC

INTERVENTIONS:
Drug: placebo for risankizumab — Placebo for risankizumab administered by intravenous infusion
  Arms: Placebo (Period 1)
Drug: risankizumab IV — Risankizumab administered by intravenous infusion
  Other Names: ABBV-066 BI 655066; SKYRIZI
  Arms: Risankizumab Dose 1 (Period 1); Risankizumab Dose 1 (Period 2); Risankizumab Dose 2 (Period 1)
Drug: risankizumab SC — Risankizumab administered by subcutaneous (SC) injection
  Other Names: ABBV-066 BI 655066; SKYRIZI
  Arms: Risankizumab Dose 2 (Period 2); Risankizumab Dose 3 (Period 2)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of risankizumab versus placebo during induction therapy in participants with moderately to severely active Crohn's disease (CD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged >=18 to <= 80 years, or minimum age of adult consent according to local regulations, at the Baseline Visit. Where locally permissible, participants 16 to < 18 years of age who meet the definition of Tanner stage 5 for development at the Baseline Visit.
* Diagnosis of CD for at least 3 months prior to Baseline.
* Confirmed diagnosis of moderate to severe CD as assessed by stool frequency (SF), abdominal pain (AP) score, and Simple Endoscopic Score for Crohn's Disease (SES-CD).
* Demonstrated intolerance or inadequate response to conventional or to biologic therapy for CD.
* If female, participant must meet the contraception recommendations.

Exclusion Criteria:

* Participant with a current diagnosis of ulcerative colitis or indeterminate colitis.
* Participants with unstable doses of concomitant Crohn's disease therapy.
* Receipt of Crohn's disease approved biologic agents (infliximab, adalimumab, certolizumab, vedolizumab, natalizumab within 8 weeks prior to Baseline or ustekinumab within 12 weeks prior to Baseline), or any investigational biologic or other agent or procedure within 35 days or 5 half-lives prior to Baseline, whichever is longer.
* Prior exposure to p19 inhibitors (e.g., risankizumab).
* Complications of Crohn's disease.
* Having an ostomy or ileoanal pouch.
* Known active Coronavirus Disease 2019 (COVID-19) infection.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 931 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2021-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (475):
- United States (117):
  - Phoenix VA Health Care System /ID# 162267, Phoenix, Arizona
  - HonorHealth Research Institute - Shea /ID# 161783, Scottsdale, Arizona
  - Digestive Disease Consultants, A Division of Arizona Digestive Health, P.C /ID# 211883, Tempe, Arizona
  - University of Arizona /ID# 158469, Tucson, Arizona
  - Atria Clinical Research /ID# 164740, Little Rock, Arkansas
  - Newport Huntington Medica /ID# 213033, Huntington Beach, California
  - United Medical Doctors /ID# 207040, Los Alamitos, California
  - TLC Clinical Research Inc /ID# 212503, Los Angeles, California
  - Gastrointestinal Biosciences Clinical Trials, LLC /ID# 162656, Los Angeles, California
  - United Medical Doctors - Murrieta /ID# 158424, Murrieta, California
  - Southern CA Research Ctr., Inc /ID# 167875, Riverside, California
  - University of California, San Francisco /ID# 157143, San Francisco, California
  - Cedars-Sinai Medical Center-West Hollywood /ID# 163842, West Hollywood, California
  - Peak Gastroenterology Associates, PC /ID# 165834, Colorado Springs, Colorado
  - Rocky Mountain Pediatric Gastroenterology /ID# 207169, Lone Tree, Colorado
  - Western Connecticut Medical Group /ID# 165849, Danbury, Connecticut
  - Seffner Premier Health Care, PA /ID# 162265, Brandon, Florida
  - Clinical Research of West Florida, Inc /ID# 204859, Clearwater, Florida
  - Clinical Research of West Florida, Inc /ID# 207450, Clearwater, Florida
  - South Lake Pain Institute, Inc /ID# 162825, Clermont, Florida
  - Universal Axon Clinical Research /ID# 165432, Doral, Florida
  - Nature Coast Clinical Research - Inverness /ID# 159414, Inverness, Florida
  - SIH Research Mumtaz, Inc /ID# 163082, Kissimmee, Florida
  - Alliance Medical Research /ID# 163840, Lighthouse PT, Florida
  - Cfagi Llc /Id# 201571, Maitland, Florida
  - Vista Health Research, LLC /ID# 212664, Miami, Florida
  - ITB Research /ID# 161334, Miami, Florida
  - Coral Research Clinic /ID# 158549, Miami, Florida
  - South Florida Research Ph I-IV, Inc. /ID# 161836, Miami, Florida
  - Gastroenterology Group Naples /ID# 165206, Naples, Florida
  - Advanced Research Institute, Inc /ID# 161959, New Port Richey, Florida
  - Endoscopic Research, Inc. /ID# 205901, Orlando, Florida
  - Omega Research Maitland, LLC /ID# 171081, Orlando, Florida
  - IMIC Inc. Medical Research /ID# 154943, Palmetto Bay, Florida
  - Clinical Research Trials of Florida, Inc. /ID# 201014, Tampa, Florida
  - Gastroenterology Associates of Central Georgia, LLC /ID# 154857, Macon, Georgia
  - Northwestern University Division of GI/Hepatology /ID# 158283, Chicago, Illinois
  - The University of Chicago Medical Center /ID# 157141, Chicago, Illinois
  - NorthShore University HealthSystem /ID# 158287, Evanston, Illinois
  - Southwest Gastroenterology /ID# 165002, Oak Lawn, Illinois
  - Cotton-O'Neil Clinical Res Ctr /ID# 154738, Topeka, Kansas
  - University of Kentucky Chandler Medical Center /ID# 157137, Lexington, Kentucky
  - University of Louisville /ID# 210521, Louisville, Kentucky
  - Gastroenterology Associates LLC - Jefferson Hwy /ID# 161956, Baton Rouge, Louisiana
  - Houma Digestive Health Special /ID# 158286, Houma, Louisiana
  - Delricht Research /ID# 206542, New Orleans, Louisiana
  - Nola Research Works, LLC /ID# 161330, New Orleans, Louisiana
  - Louisana Research Center, LLC /ID# 162236, Shreveport, Louisiana
  - MGG Group Co, Inc.Chevy Chase Clinical Research /ID# 154839, Chevy Chase, Maryland
  - Gastro Center of Maryland /ID# 165004, Columbia, Maryland
  - University of Michigan Health Systems /ID# 157144, Ann Arbor, Michigan
  - Center for Digestive Health /ID# 154690, Troy, Michigan
  - Gastroenterology Associates of Western Michigan, PLC d.b.a. West Michigan Clinic /ID# 161328, Wyoming, Michigan
  - Mayo Clinic - Rochester /ID# 163085, Rochester, Minnesota
  - Southern Therapy and Advanced Research (STAR) LLC /ID# 162388, Jackson, Mississippi
  - St. Louis University /ID# 161902, St Louis, Missouri
  - University of Nebraska Medical Center /ID# 210057, Omaha, Nebraska
  - Las Vegas Medical Research /ID# 160172, Las Vegas, Nevada
  - Revival Research Institute, Inc /ID# 210984, Las Vegas, Nevada
  - NY Scientific /ID# 158418, Brooklyn, New York
  - Saratoga Schenectady Gastroenterology Associates - Burnt Hills /ID# 212036, Burnt Hills, New York
  - Intercity Advanced Gastroentertology Center /ID# 213399, Fresh Meadows, New York
  - Duplicate_Long Island Clinical Research /ID# 154836, Great Neck, New York
  - Digestive Disease Care /ID# 209619, New Hyde Park, New York
  - North Shore University Hospital /ID# 168736, New Hyde Park, New York
  - NYU Langone Medical Center /ID# 160171, New York, New York
  - Columbia Univ Medical Center /ID# 161911, New York, New York
  - Lenox Hill Hospital /ID# 168465, New York, New York
  - DiGiovanna Institute for Medical Education & Research /ID# 171118, North Massapequa, New York
  - Univ NC Chapel Hill /ID# 154840, Chapel Hill, North Carolina
  - Atrium Health Carolinas Medical Center /ID# 158481, Charlotte, North Carolina
  - Clinical Trials America /ID# 158484, Hickory, North Carolina
  - Vidant Multispecialty Clinic - Kinston /ID# 161111, Kinston, North Carolina
  - Wake Radiology UNC REX Healthcare - Raleigh Office /ID# 154880, Raleigh, North Carolina
  - Plains Clinical Research Center, LLC /ID# 169715, Fargo, North Dakota
  - Tri-State Endoscopy /ID# 154933, Cincinnati, Ohio
  - Cleveland Clinic Main Campus /ID# 208171, Cleveland, Ohio
  - The Ohio State University /ID# 164709, Columbus, Ohio
  - Optimed Research, Ltd. /ID# 167901, Columbus, Ohio
  - Hometown Urgent Care and Resea /ID# 170453, Dayton, Ohio
  - Great Lakes Medical Research, LLC /ID# 201732, Mentor, Ohio
  - Hightower Clinical /ID# 211938, Oklahoma City, Oklahoma
  - Digestive Disease Specialists /ID# 170774, Oklahoma City, Oklahoma
  - Adult Gastroenterology Associates - Gen 1 Research /ID# 206125, Tulsa, Oklahoma
  - Northwest Gastroenterology Clinic /ID# 158288, Portland, Oregon
  - PennState Milton S.Hershey Med /ID# 154883, Hershey, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC /ID# 210920, Pittsburgh, Pennsylvania
  - Digestive Disease Associates, LTD /ID# 208847, Wyomissing, Pennsylvania
  - Medical University of South Carolina /ID# 212579, Charleston, South Carolina
  - Gastroenterology Associates, P.A. of Greenville /ID# 154911, Greenville, South Carolina
  - Rapid City Medical Center - GI Research /ID# 163841, Rapid City, South Dakota
  - Gastro One /ID# 154742, Germantown, Tennessee
  - East Tennessee Research Institute /ID# 168737, Johnson City, Tennessee
  - Duplicate_Clinical Neuroscience Solutions /ID# 164181, Memphis, Tennessee
  - Vanderbilt University Medical Center /ID# 157138, Nashville, Tennessee
  - TX Clinical Research Institute /ID# 159410, Arlington, Texas
  - Inquest Clinical Research /ID# 165695, Baytown, Texas
  - Texas Digestive Disease Consultants /ID# 209596, Cedar Park, Texas
  - Texas Digestive Disease Consultants /ID# 209785, Cedar Park, Texas
  - Baylor Scott & White Center for Inflammatory Bowel Diseases /ID# 201848, Dallas, Texas
  - DHAT Research Institute /ID# 158217, Garland, Texas
  - Vilo Research Group Inc /ID# 206130, Houston, Texas
  - CliniCore International, LLC /ID# 158209, Houston, Texas
  - Baylor College of Medicine - Baylor Medical Center /ID# 158212, Houston, Texas
  - Precision Research Institute, LLC /ID# 200503, Houston, Texas
  - Centex Studies, Inc. - Houston /ID# 200720, Houston, Texas
  - Clinical Associates in Research Therapeutics of America, LLC /ID# 161336, San Antonio, Texas
  - Southern Star Research Institute, LLC /ID# 168770, San Antonio, Texas
  - Tyler Research Institute, LLC /ID# 166796, Tyler, Texas
  - Gastro Health & Nutrition - Victoria /ID# 164296, Victoria, Texas
  - HP Clinical Research /ID# 162998, Bountiful, Utah
  - Advanced Research Institute /ID# 154914, Ogden, Utah
  - Velocity Clinical Research - Salt Lake City /ID# 161781, West Jordan, Utah
  - McGuire DV AMC /ID# 159990, Richmond, Virginia
  - Washington Gastroenterology Associates /ID# 162120, Bellevue, Washington
  - Virginia Mason - Seattle Orthapedics /ID# 155545, Seattle, Washington
  - WVU Medicine /ID# 167940, Morgantown, West Virginia
- Argentina (2):
  - Duplicate_HOSPITAL CENTENARIO /ID# 170883, Rosario, Santa Fe Province
  - Hospital Privado Univesitario /ID# 161988, Córdoba
- Australia (5):
  - Duplicate_Mater Hospital /ID# 167990, South Brisbane, Queensland
  - Griffith University /ID# 212627, Southport, Queensland
  - Lyell McEwin Hospital /ID# 211363, Elizabeth Vale, South Australia
  - Emeritus Research /ID# 213511, Camberwell, Victoria
  - Footscray Hospital /ID# 211361, Footscray, Victoria
- Austria (4):
  - Universitaetsklinikum St. Poelten /ID# 166425, Sankt Pölten, Lower Austria
  - Medizinische Universitaet Graz /ID# 158137, Graz, Styria
  - Krankenhaus der Barmherzigen Brueder Wien /ID# 212059, Vienna, Vienna
  - Duplicate_Medical University of Vienna /ID# 158138, Vienna, Vienna
- Belarus (3):
  - Grodno city clinical hospital #2 /ID# 159499, Grodno
  - Gomel Regional Clinical Hospital /ID# 159498, Homyel
  - Vitebsk Regional Advanced Clin /ID# 159497, Vitebsk
- Belgium (9):
  - ULB Hospital Erasme /ID# 157397, Brussels, Brussels Capital
  - UCL Saint-Luc /ID# 157395, Woluwe-Saint-Lambert, Brussels Capital
  - CHU UCL Namur - site Godinne /ID# 157401, Godinne, Namur
  - UZ Gent /ID# 157394, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 157396, Leuven, Vlaams-Brabant
  - Imelda Ziekenhuis /ID# 157392, Bonheiden
  - CHU de Liege /ID# 157398, Liège
  - Groupe Sante CHC - Clinique du MontLegia /ID# 157393, Liège
  - AZ-Delta /ID# 157391, Roeselare
- Bosnia and Herzegovina (3):
  - University Clinical Centre of the Republic of Srpska /ID# 157717, Banja Luka, Republika Srpska
  - University Clinical Centre of the Republic of Srpska /ID# 164512, Banja Luka, Republika Srpska
  - Clinical Center University of Sarajevo /ID# 165134, Sarajevo
- Brazil (7):
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva /ID# 157672, Goiânia, Goiás
  - Hospital Nossa Senhora das Graças /ID# 157646, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre /ID# 157653, Porto Alegre, Rio Grande do Sul
  - Upeclin Fmb - Unesp /Id# 157688, Botucatu, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto - USP /ID# 157649, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC /ID# 159672, Santo André, São Paulo
  - Kaiser Clinica e Hospital Dia /ID# 157656, São José do Rio Preto, São Paulo
- Bulgaria (8):
  - UMHAT Dr Georgi Stranski EAD /ID# 203977, Pleven
  - University Multiprofile Hospit /ID# 158644, Plovdiv
  - Second Multiprofile Hospital f /ID# 158646, Sofia
  - Duplicate_Tokuda Hospital Sofia /ID# 158645, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 204714, Sofia
  - UMHAT Tsaritsa Joanna - ISUL /ID# 211240, Sofia
  - MHAT Trakia /ID# 201672, Stara Zagora
  - University Multiprofile Hospit /ID# 167575, Varna
- Canada (19):
  - University of Calgary - Heritage Medical Research Clinic /ID# 157152, Calgary, Alberta
  - Allen Whey Khye Lim Professional Corporation /ID# 169761, Edmonton, Alberta
  - University of Alberta - Zeidler Ledcor Centre /ID# 157098, Edmonton, Alberta
  - Covenant Health /ID# 161617, Edmonton, Alberta
  - Fraser Clinical Trials Inc /ID# 159053, New Westminster, British Columbia
  - GIRI Gastrointestinal Research Institute /ID# 157095, Vancouver, British Columbia
  - Percuro Clinical Research, Ltd /ID# 161616, Victoria, British Columbia
  - QEII - Health Sciences Centre /ID# 157087, Halifax, Nova Scotia
  - IWK Health Center /ID# 165900, Halifax, Nova Scotia
  - Medicor Research Inc /ID# 157149, Greater Sudbury, Ontario
  - London Health Sciences Center /ID# 157160, London, Ontario
  - Scott Shulman Medicine Professional Corporation /ID# 165903, North Bay, Ontario
  - Mount Sinai Hospital /ID# 169762, Toronto, Ontario
  - Toronto Digestive Disease Asso /ID# 157157, Vaughan, Ontario
  - CISSS de la Monteregie /ID# 161615, Greenfield Park, Quebec
  - CHAU- Hotel-Dieu de Levis /ID# 214375, Lévis, Quebec
  - CIUSSS de l'est de l'Ile-de-Montreal - Hopital Maisonneuve-Rosemont /ID# 159054, Montreal, Quebec
  - CHUM - Centre hospitalier de l'Universite de Montréal /ID# 167066, Montreal, Quebec
  - Montreal General Hospital - McGill University Health Center /ID# 157084, Montreal, Quebec
- Chile (4):
  - Centro de Investigaciones Clínicas Viña del Mar /ID# 203589, Viña del Mar, Región de Valparaíso
  - Complejo Asistencial Dr. Sotero del Rio /ID# 169382, Santiago, Santiago Metropolitan
  - Hospital Guillermo Grant Benavente de Concepción /ID# 210759, Concepción
  - Hospital Las Higueras /ID# 167090, Talcahuano
- China (16):
  - Guangdong Provincial People's Hospital /ID# 212948, Guangzhou, Guangdong
  - The Sixth Affiliated Hosp Sun /ID# 210785, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University /ID# 212740, Shijiazhuang, Hebei
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Techno /ID# 210856, Wuhan, Hubei
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Sc /ID# 211038, Wuhan, Hubei
  - Renmin Hospital of Wuhan University /ID# 214873, Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University /ID# 211034, Nanchang, Jiangxi
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 210841, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine /ID# 210707, Shanghai, Shanghai Municipality
  - The second Affiliated hospital of Zhejiang University school of Medicine /ID# 210725, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine /ID# 210624, Hangzhou, Zhejiang
  - Jinhua Municipal Central Hospital /ID# 215626, Jinhua, Zhejiang
  - The Second Hospital Central South University /ID# 211696, Changsha
  - West China Hospital, Sichuan University /ID# 210889, Chengdu
  - Shanghai East Hospital /ID# 212683, Pudong New District
  - Tianjin Medical University General Hospital /ID# 210927, Tianjin
- Colombia (4):
  - Instituto de Coloproctologia /ID# 158741, Medellín, Antioquia
  - Hospital Pablo Tobon Uribe /ID# 158735, Medellín, Antioquia
  - Hospital Univ San Ignacio /ID# 158733, Bogota, Cundinamarca
  - Hospital Universitario San Vic /ID# 171487, Medellín
- Croatia (5):
  - Duplicate_Klinicka bolnica Dubrava Zagreb /ID# 157565, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Sestre milosrdnice /ID# 157721, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 157566, Zagreb, City of Zagreb
  - UHC Osijek /ID# 157564, Osijek, County of Osijek-Baranja
  - Klinicki bolnicki centar Split /ID# 157567, Split, Split-Dalmatia County
- Czechia (9):
  - Duplicate_Institut klinicke a experimentalni mediciny (IKEM) /ID# 165463, Prague, Praha 4
  - Hepato-Gastroenterologie HK, s.r.o. /ID# 163134, Hradec Králové
  - CTCenter MaVe s.r.o. /ID# 163149, Olomouc
  - Nemocnice Pardubickeho kraje, a.s. /ID# 163182, Pardubice
  - Nemocnice Milosrdnych sester sv. Karla Boromejskeho v Praze /ID# 211305, Prague
  - Axon Clinical, s.r.o. /ID# 163176, Prague
  - Thomayerova nemocnice /ID# 162940, Prague
  - ResTrial s.r.o. /ID# 211075, Prague
  - NH Hospital a.s. /ID# 211076, Prague
- Estonia (3):
  - East Tallinn Central Hospital /ID# 157076, Tallinn, Harju
  - West Tallinn Central Hospital /ID# 157077, Tallinn
  - North Estonia Medical Centre /ID# 163507, Tallinn
- Germany (31):
  - Universitaetsklinikum Freiburg /ID# 162019, Freiburg im Breisgau, Baden-Wurttemberg
  - Praxis fuer Gastroenterologie /ID# 166145, Heidelberg, Baden-Wurttemberg
  - Universitatsklinikum Mannheim /ID# 162020, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen /ID# 159324, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 164986, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 159315, Erlangen, Bavaria
  - Universitaetsklinikum Frankfurt /ID# 212978, Frankfurt am Main, Hesse
  - Universitaetsklinikum Koeln /ID# 164985, Cologne, North Rhine-Westphalia
  - Evangelisches Krankenhaus Kalk /ID# 212725, Cologne, North Rhine-Westphalia
  - Praxiszentrum fuer Gastroenterologie /ID# 211964, Grevenbroich, North Rhine-Westphalia
  - Universitaetsklinikum Muenster /ID# 159316, Münster, North Rhine-Westphalia
  - Zentrum für Gastroenterologie Saar MVZ GmbH /ID# 210529, Saarbrücken, Saarland
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 159321, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Jena /ID# 159323, Jena, Thuringia
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 212219, Berlin
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 212893, Berlin
  - Gastroenterologische Spezialpraxis am Wittenbergplatz /ID# 211972, Berlin
  - MVZ fuer Gastroenterlogie am Bayerischen Platz /ID# 159322, Berlin
  - DRK Kliniken Berlin Westend /ID# 166146, Berlin
  - Krankenhaus Waldfriede /ID# 212728, Berlin-Zehlendorf
  - Stadtisches Klinikum Braunschweig /ID# 163666, Braunschweig
  - Medizinisches Versorgunszentrum Dachau /ID# 211557, Dachau
  - Agaplesion Markus Krankenhaus /ID# 159317, Frankfurt am Main
  - Asklepios Westklinikum Hamburg /ID# 159319, Hamburg
  - Medizinische Hochschule Hannover /ID# 162021, Hanover
  - EUGASTRO GmbH /ID# 212076, Leipzig
  - Klinikum Lueneburg /ID# 163664, Lüneburg
  - Universitaetsklinikum Magdeburg /ID# 211847, Magdeburg
  - Gastroenterologische Gemeinschaftspraxis Minden /ID# 162018, Minden
  - Universitaetsklinikum Regensburg /ID# 163665, Regensburg
  - Duplicate_Gastro-Praxis Wiesbaden /ID# 159318, Wiesbaden
- Greece (7):
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 171077, Athens, Attica
  - Tzaneio general hospital of Piraeus /ID# 206445, Piraeus, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 157427, Heraklion, Crete
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 157428, Athens
  - University General Hospital of Ioannina /ID# 157425, Ioannina
  - General Hospital of Nikaia-Piraeus "Agios Panteleimon"- general hospital dytikis /ID# 157429, Pireaus
  - Theageneio Anticancer Hospital /ID# 163921, Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital /ID# 163902, Hong Kong
  - Tuen Mun Hospital /ID# 163901, Tuenmen
- Ireland (3):
  - Beaumont Hospital /ID# 157515, Beaumont, Dublin
  - St Vincent's University Hospital /ID# 157512, Elm Park, Dublin
  - University Hospital Galway /ID# 157513, Galway
- Israel (9):
  - Soroka University Medical Center /ID# 157798, Beersheba, Southern District
  - Sheba Medical Center /ID# 157797, Ramat Gan, Tel Aviv
  - Sheba Medical Center /ID# 171074, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 157796, Tel Aviv, Tel Aviv
  - Duplicate_Rambam Medical Center /ID# 171072, Haifa
  - The Edith Wolfson Medical Center /ID# 217329, Holon
  - Shaare Zedek Medical Center /ID# 163540, Jerusalem
  - Shaare Zedek Medical Center /ID# 171073, Jerusalem
  - Hadassah Medical Center-Hebrew University /ID# 165913, Jerusalem
- Italy (18):
  - Duplicate_AOU Ospendali Riuniti di Ancona /ID# 162427, Torrette, Ancona
  - University of Catanzaro /ID# 212012, Catanzaro, Calabria
  - Duplicate_Azienda Ospedaliero-Universitaria Policlinico di Modena /ID# 212019, Modena, Emilia-Romagna
  - Policlinico Universitario Campus Bio-Medico /ID# 162429, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini /ID# 155636, Rome, Lazio
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 166911, Rome, Lazio
  - Istituto Clinico Humanitas /ID# 155634, Rozzano, Milano
  - Fondazione PTV Policlinico Tor Vergata /ID# 158021, Rome, Roma
  - Presidio Columbus-Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Un /ID# 155632, Rome, Roma
  - Duplicate_Azienda Ospedaliera Univ. Meyer /ID# 168051, Florence, Tuscany
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 161305, Negrar, Verona
  - A.O.U. di Bologna Policlinico S.Orsola-Malpighi /ID# 155635, Bologna
  - A.O. Per L'Emergenza Cannizzaro /ID# 161306, Catania
  - Ospedale Policlinico San Martino /ID# 162430, Genova
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 155633, Milan
  - ASST Fatebenefratelli Sacco-Ospedale Sacco /ID# 155631, Milan
  - A.O. Ospedali Riuniti Villa Sofia - Cervello /ID# 155637, Palermo
  - Duplicate_Fondazione IRCCS Policlinico San Matteo /ID# 212029, Pavia
- Japan (45):
  - Aichi Medical University Hospital /ID# 160159, Nagakute-shi, Aichi-ken
  - Daido Clinic /ID# 211477, Nagoya, Aichi-ken
  - Nagoya University Hospital /ID# 160150, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 160162, Nagoya, Aichi-ken
  - Fujita Health University Hospital /ID# 163214, Toyoake-shi, Aichi-ken
  - Tokatsu Tsujinaka Hospital /ID# 163362, Abiko-shi, Chiba
  - Chiba University Hospital /ID# 217532, Chiba, Chiba
  - Tsujinaka Hospital Kashiwanoha /ID# 213847, Kashiwa-shi, Chiba
  - The Jikei University Kashiwa Hospital /ID# 200007, Kashiwa-shi, Chiba
  - Toho University Sakura Medical Center /ID# 160161, Sakura-shi, Chiba
  - Fukuoka University Hospital /ID# 217792, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 160138, Kurume-shi, Fukuoka
  - NHO Fukuyama Medical Center /ID# 163578, Fukuyama-shi, Hiroshima
  - Hiroshima University Hospital /ID# 160139, Hiroshima, Hiroshima
  - Asahikawa Medical University Hospital /ID# 162844, Midorigaokahiga-shi, Hokkaido
  - Sapporo Tokushukai Hospital /ID# 213493, Sapporo, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 160158, Sapporo, Hokkaido
  - Sapporo Medical University Hospital /ID# 163028, Sapporo, Hokkaido
  - Nishinomiya Munic Central Hospital /ID# 210104, Nishinomiya-shi, Hyōgo
  - Hyogo College of Medicine College Hospital /Id# 160164, Nishinomiya-shi, Hyōgo
  - National Hospital Organization Mito Medical Center /ID# 160154, Higashi Ibaraki-gun, Ibaraki
  - Kanazawa University Hospital /ID# 201766, Kanazawa, Ishikawa-ken
  - Gokeikai Ofuna Chuo Hospital /ID# 171070, Kamakura-shi, Kanagawa
  - Kitasato University Hospital /ID# 171071, Sagamihara-shi, Kanagawa
  - Yokohama City University Medical Center /ID# 163906, Yokohama, Kanagawa
  - Yokohama Municipal Citizen's Hospital /ID# 204126, Yokohama, Kanagawa
  - Mie University Hospital /ID# 203639, Tsu, Mie-ken
  - Yokkaichi Hazu Medical Center /ID# 163741, Yokkaichi-shi, Mie-ken
  - Tohoku University Hospital /ID# 162843, Sendai, Miyagi
  - Duplicate_Tohoku Rosai Hospital /ID# 163189, Sendai, Miyagi
  - Osaka City University Hospital /ID# 160146, Osaka, Osaka
  - Saitama Medical Center /ID# 160155, Kawagoe-shi, Saitama
  - Tokitokai Tokito clinic /ID# 160145, Saitama-shi, Saitama
  - Shiga University of Medical Science Hospital /ID# 164022, Ōtsu, Shiga
  - Hamamatsu University Hospital /ID# 205689, Hamamatsu, Shizuoka
  - NHO Shizuoka Medical Center /ID# 163029, Sunto-gun, Shizuoka
  - Tokyo Medical And Dental University, Medical Hospital /ID# 160157, Bunkyo-ku, Tokyo
  - Duplicate_Tokai University Hachioji Hospital /ID# 160160, Hachioji-shi, Tokyo
  - The Jikei University Hospital /ID# 163190, Minato-ku, Tokyo
  - Duplicate_Kitasato University Kitasato Institute Hospital /ID# 160144, Minato-ku, Tokyo
  - Kyorin University Hospital /ID# 160149, Mitaka-shi, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 205973, Shinjuku-ku, Tokyo
  - Wakayama Medical University Hospital /ID# 200183, Wakayama, Wakayama
  - Yamagata University Hospital /ID# 200154, Yamagata, Yamagata
  - Yamanashi Prefectural Central Hospital /ID# 160156, Kofu, Yamanashi
- Latvia (3):
  - Pauls Stradins Clinical University Hospital /ID# 159614, Riga
  - Digestive Disease Center Gastro /ID# 163105, Riga
  - Riga East Clinical University Hospital /ID# 159613, Riga
- Lithuania (2):
  - Duplicate_Hospital of lithuanian university of Health Science Kauno Klinikos /ID# 162582, Kaunas
  - Duplicate_Vilnius University Hospital /ID# 162507, Vilnius
- Malaysia (3):
  - Universiti Sains Malaysia /ID# 160656, Kelantan, Kelantan
  - Queen Elizabeth Hospital /ID# 160654, Division Pantai Barat Utara, Sabah
  - Universiti Kebangsaan Malaysia (UKM) Medical Centre /ID# 163654, Kuala Lumpur, Selangor
- Mexico (4):
  - Investigacion Biomedica para el Desarrollo de Farmacos, S.A. de C.V. /ID# 167648, Zapopan, Jalisco
  - JM Research SC /ID# 161733, Cuernavaca, Morelos
  - Unidad de Atencion Medica e Investigacion en Salud /ID# 163624, Mérida, Yucatán
  - Health Pharma Professional Research S.A de C.V /ID# 161734, Del. Benito Juárez
- Netherlands (2):
  - Academisch Medisch Centrum /ID# 157950, Amsterdam
  - Elisabeth Tweesteden Ziekenhuis /ID# 163631, Tilburg
- New Zealand (3):
  - Christchurch Hospital /ID# 163074, Christchurch, Canterbury
  - Dunedin Hospital /ID# 167989, Dunedin, Otago
  - Wellington Regional Hospital /ID# 167987, Newtown Wellington, Wellington Region
- Norway (4):
  - Akershus universitetssykehus /ID# 169378, Nordbyhagen, Akershus
  - Helse More og Romsdal HF, Alesund sjukehus /ID# 212811, Ålesund
  - Vestre viken - Baerum Sykehus /ID# 157886, Gjettum
  - Sykehuset Levanger Helse NT /ID# 157885, Levanger
- Poland (15):
  - Gastromed /Id# 212099, Torun, Kuyavian-Pomeranian Voivodeship
  - Planetmed Sp. z o.o. /ID# 202798, Wroclaw, Lower Silesian Voivodeship
  - 1 Wojskowy Szpital Kliniczny Z Poliklinika /Id# 209985, Lublin, Lublin Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie /ID# 209981, Lublin, Lublin Voivodeship
  - Centrum Zdrowia MDM /ID# 160794, Warsaw, Masovian Voivodeship
  - Centralny Szpital Kliniczny MSWiA w Warszawie /ID# 160797, Warsaw, Masovian Voivodeship
  - Instytut Pomnik - Centrum Zdrowia Dziecka /ID# 213579, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Medyk /ID# 212889, Rzeszów, Podkarpackie Voivodeship
  - Centrum Medyczne LukaMed Joanna Luka-Wendrowska /ID# 212081, Chojnice, Pomeranian Voivodeship
  - H-T. Centrum Medyczne - Endoterapia /ID# 212459, Tychy, Silesian Voivodeship
  - Wojewodzki Szpital Specjalistyczny /ID# 212402, Olsztyn, Warmian-Masurian Voivodeship
  - Duplicate_SOLUMED Sp. z o.o., Sp.k. /ID# 160793, Poznan
  - Duplicate_Niepubliczny Zakład Opieki Zdrowotnej VIVAMED Jadwiga Miecz /ID# 205160, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclaw /ID# 212602, Wroclaw
  - Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego w Lodzi /ID# 212297, Lodz, Łódź Voivodeship
- Portugal (11):
  - Hospital da Senhora da Oliveira Guimaraes, EPE /ID# 160739, Guimarães, Braga District
  - Centro Hospitalar Universitário do Algarve, EPE - Hospital de Portimão /ID# 167750, Portimão, Faro District
  - Centro Hospitalar de Entre Douro e Vouga /ID# 160674, Santa Maria DA Feira, Porto District
  - Hospital Garcia de Orta, EPE /ID# 160747, Almada
  - Centro Hospitalar Universitário do Algarve, EPE - Hospital Faro /ID# 160715, Faro
  - Centro Hospitalar Universitario Lisboa Central, EPE - Hospital dos Capuchos /ID# 160675, Lisbon
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital Egas Moniz /ID# 167749, Lisbon
  - Centro Hospitalar Universitário de Lisboa Norte, EPE - Hospital de Santa Maria /ID# 160694, Lisbon
  - Hospital Beatriz Ângelo /ID# 207757, Loures
  - Centro Hospitalar Universitario de Sao Joao, EPE /ID# 160695, Porto
  - Centro Hosp de Tondela-Viseu /ID# 160697, Viseu
- Romania (5):
  - Institutul Clinic Fundeni /ID# 163046, Sector 2, București
  - Institutul Clinic Fundeni /ID# 163264, Sector 2, București
  - Tvm Med Serv Srl /Id# 166294, Cluj-Napoca
  - Cabinet Particular Policlinic Algomed /ID# 163047, Timișoara
  - Duplicate_Centrul Medical Tuculanu SRL /ID# 166295, Timișoara
- Russia (11):
  - Kuzbass Regional Clinical Hospital /ID# 161310, Kemerovo, Kemerovo Oblast
  - Duplicate_Perm state medical university n.a. E.A. Vagner /ID# 207440, Perm, Permskiy Kray
  - Duplicate_St. Petersburg State Pediatric Medical University /ID# 211977, Saint Petersburg, Sankt-Peterburg
  - Professor Pasechnikov Gastroenterology and Pankreatology clinic /ID# 156949, Stavropol, Stavropol Kray
  - Tver Regional Clinical Hospital /ID# 205925, Tver', Tver Oblast
  - Regional Clinical Hospital #1 /ID# 163453, Tyumen, Tyumen Oblast
  - Alliance Biomedical Ural Group /ID# 156950, Izhevsk, Udmurtiya Republic
  - State Scientific Ctr Coloproct /ID# 204809, Moscow
  - Novosibirski Gastrocenter /ID# 217554, Novosibirsk
  - City Clinical Hospital No. 31 /ID# 208866, Saint Petersburg
  - Duplicate_Ulyanovsk State clinical hospi /ID# 156946, Ulyanovsk
- Serbia (9):
  - Clinical Hosp Center Zvezdara /ID# 156978, Belgrade, Beograd
  - Military Medical Academy /ID# 156979, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 156973, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 156976, Belgrade, Beograd
  - University Clinical Center Kragujevac /ID# 156975, Kragujevac, Sumadijski Okrug
  - Clinical Center Vojvodina /ID# 156972, Novi Sad, Vojvodina
  - University Children's Hospital 'Tirsova' /ID# 211481, Belgrade
  - Clinical Hospital Center Dr Dragisa Misovic - Dedinje /ID# 212797, Belgrade
  - General Hospital Leskovac /ID# 209574, Leskovac
- Singapore (3):
  - National University Hospital /ID# 160658, Singapore
  - Singapore General Hospital /ID# 160657, Singapore
  - KL Ling Gastroenterology and Liver Clinic /ID# 205737, Singapore
- Slovakia (4):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 156465, Banská Bystrica
  - Univerzitna nemocnica Martin /ID# 163200, Martin
  - KM Management, spol. s.r.o. /ID# 206763, Nitra
  - GASTRO I., s.r.o. /ID# 156466, Prešov
- South Africa (5):
  - Clinresco Centers /ID# 163864, Johannesburg, Gauteng
  - Wits Clinical Research Site /ID# 158115, Johannesburg, Gauteng
  - Kingsbury Hospital /ID# 163116, Cape Town, Western Cape
  - Private Practice Dr MN Rajabally /ID# 163115, Cape Town, Western Cape
  - Spoke Research Inc /ID# 158117, CAPE TOWN Milnerton, Western Cape
- South Korea (11):
  - Hanyang University Guri Hospital /ID# 158673, Guri-si, Gyeonggido
  - Duplicate_CHA bundang medical center CHA University /ID# 158672, Seongnam-si, Gyeonggido
  - Duplicate_The Catholic University of Korea, ST. Vincent's Hospital /ID# 158681, Suwon, Gyeonggido
  - Kangbuk Samsung Hospital /ID# 158676, Seoul, Seoul Teugbyeolsi
  - Severance Hospital /ID# 158671, Seoul, Seoul Teugbyeolsi
  - Dong-A University Hospital /ID# 158675, Busan
  - Pusan National University Hospital /ID# 158677, Busan
  - Yeungnam University Medical Center /ID# 158680, Daegu
  - The Catholic University of Korea, Daejeon St.Mary's Hospital /ID# 213552, Daejeon
  - Asan Medical Center /ID# 158678, Seoul
  - Samsung Medical Center /ID# 158674, Seoul
- Spain (12):
  - Hospital Arquitecto Marcide - Complejo Hospitalario Universitario de Ferrol /ID# 157527, Ferrol, A Coruna
  - Consorci Corporacio Sanitaria Parc Tauli Sabadell /ID# 159230, Sabadell, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda /ID# 157575, Majadahonda, Madrid
  - Hospital Universitario Basurto /ID# 205189, Bilbao, Vizcaya
  - Hospital Clinic de Barcelona /ID# 157526, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 161435, Madrid
  - Hospital Universitario La Paz /ID# 159228, Madrid
  - Hospital Clinico Universitario de Salamanca /ID# 157532, Salamanca
  - Hospital Universitario Virgen Macarena /ID# 160819, Seville
  - Hospital Universitario y Politecnico La Fe /ID# 157530, Valencia
  - Hospital Clinico Universitario Lozano Blesa /ID# 212523, Zaragoza
  - Hospital Universitario Miguel Servet /ID# 157531, Zaragoza
- Sweden (7):
  - Skane University hospital /ID# 211235, Malmo, Skåne County
  - Duplicate_GHP Stockholm Gastro Center /ID# 210479, Stockholm, Stockholm County
  - Ersta diakoni /ID# 157878, Stockholm, Stockholm County
  - Danderyd Hospital /ID# 202136, Stockholm, Stockholm County
  - Sahlgrenska University Hospital /ID# 157879, Gothenburg, Västra Götaland County
  - Duplicate_SU Molndal. /ID# 157880, Mölndal
  - Duplicate_Karolinska Univ Sjukhuset /ID# 209966, Solna
- Switzerland (3):
  - Universitätsspital Zürich /ID# 163532, Zurich, Canton of Zurich
  - Duplicate_Universitaetsspital Basel /ID# 164555, Basel
  - Inselspital, Universitätsspital Bern /ID# 163531, Bern
- Ukraine (12):
  - Scientific Research Institute of Invalid Rehabilitation /ID# 211516, Vinnytsia, Vinnytsia Oblast
  - Kharkiv City Clinical Hospital No.2 n.a. Prof. O.O. Shalimov /ID# 165649, Kharkiv
  - Municipal Nonprofit Enterprise Kherson city clinical hospital n.a. Y.Y. Karabel /ID# 212050, Kherson
  - Kyiv Municipal Clinical Hospital #18 /ID# 162521, Kyiv
  - International Institute of Clinical Research LLC /ID# 211997, Kyiv
  - Communal Noncommercial Institution Consultative and Diagnostic Center of Desnian /ID# 165651, Kyiv
  - Medical Center of LLC Medbud-Clinic /ID# 216929, Kyiv
  - Kyiv Railway Clinical Hosp No.2 /ID# 217330, Kyiv
  - Communal Enterprise Volyn Regional Clinical hospital of the Volyn Regional Coun /ID# 206788, Lutsk
  - Lviv Railway Clinical Hospital of branch Healthcare Centers of Public Joint Stoc /ID# 165650, Lviv
  - Duplicate_Transcarpathian Regional Clin. /ID# 168419, Uzhhorod
  - MNPE Vinnytsia Regional Clinical Hospital n.a. M.I. Pyrohov /ID# 216265, Vinnytsia
- United Kingdom (13):
  - Royal Devon and Exeter NHS Trust Hospital /ID# 157517, Exeter, Devon
  - Barts Health NHS Trust /ID# 163710, London, London, City of
  - Guy's and St Thomas' NHS Foundation Trust /ID# 157519, London, London, City of
  - Ashford and St Peter's Hospitals NHS Foundation Trust /ID# 207937, Chertsey, Surrey
  - Cambridge University Hospitals NHS Foundation Trust /ID# 158031, Cambridge
  - NHS Lothian /ID# 207447, Edinburgh
  - Calderdale and Huddersfield NHS Foundation Trust /ID# 209569, Huddersfield
  - Hull University Teaching Hospitals NHS Trust /ID# 158757, Hull
  - Leeds Teaching Hospitals NHS Trust /ID# 157523, Leeds
  - Duplicate_King's College Hospital NHS Foundation Trusts /ID# 158756, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 163709, Newcastle upon Tyne
  - Oxford University Hospitals NHS Foundation Trust /ID# 158033, Oxford
  - Duplicate_Northern Care Alliance NHS Group /ID# 207764, Salford

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Panaccione R, Ferrante M, Dotan I, Panes J, Hisamatsu T, Bossuyt P, Danese S, Song A, Kalabic J, Joshi N, Zambrano J, Zhang Y, Duan WR, Kligys K, Dubinsky MC, Lindsay JO, Vermeire S, Siegmund B, Irving PM, D'Haens G. Extended Risankizumab Treatment in Patients With Crohn's Disease Who Did Not Achieve Clinical Response to Induction Treatment. Clin Gastroenterol Hepatol. 2025 Oct;23(11):2012-2022.e6. doi: 10.1016/j.cgh.2024.12.023. Epub 2025 Feb 3. PMID 39909280
- [Derived] Atreya R, Ferrante M, Panaccione R, Feagan B, Shchukina O, Jairath V, Rieder F, Hisamatsu T, Siegmund B, Kligys K, Song A, Zambrano J, Mallick M, Zhang Y, Armuzzi A, D'Haens G. Risankizumab Is Associated With Normalization of Biomarkers in Patients With Crohn's Disease: Results From the Phase 3 ADVANCE, MOTIVATE, and FORTIFY Studies. J Crohns Colitis. 2025 Apr 4;19(4):jjae164. doi: 10.1093/ecco-jcc/jjae164. PMID 39485390
- [Derived] Peyrin-Biroulet L, Colombel JF, Louis E, Ferrante M, Motoya S, Panaccione R, Torres J, Ungaro RC, Kligys K, Kalabic J, Zambrano J, Zhang Y, D'Haens G. Shorter Crohn's Disease Duration Is Associated With Better Clinical and Endoscopic Outcomes With Risankizumab in Phase 3 Studies. Gastro Hep Adv. 2024 Mar 7;3(4):539-550. doi: 10.1016/j.gastha.2024.02.008. eCollection 2024. PMID 39131711
- [Derived] Louis E, Lee WJ, Litcher-Kelly L, Ollis S, Pranschke E, Fitzgerald K, Lacerda AP, Neimark E, Sanchez Gonzalez Y, Panes J. Content Validity and Psychometric Evaluation of the Crohn's Symptom Severity (CSS) Questionnaire in Patients with Moderately to Severely Active Crohn's Disease. Adv Ther. 2024 Sep;41(9):3678-3705. doi: 10.1007/s12325-024-02923-9. Epub 2024 Aug 6. PMID 39105965
- [Derived] Dubinsky M, Ma C, Griffith J, Crowell M, Neimark E, Kligys K, O'Connell T. Matching-Adjusted Indirect Comparison Between Risankizumab and Ustekinumab for Induction and Maintenance Treatment of Moderately to Severely Active Crohn's Disease. Adv Ther. 2023 Sep;40(9):3896-3911. doi: 10.1007/s12325-023-02546-6. Epub 2023 Jun 27. PMID 37368103
- [Derived] Loftus EV Jr, Ananthakrishnan AN, Lee WJ, Gonzalez YS, Fitzgerald KA, Wallace K, Zhou W, Litcher-Kelly L, Ollis SB, Su S, Danese S. Content Validity and Psychometric Evaluation of the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) in Patients with Crohn's Disease and Ulcerative Colitis. Pharmacoecon Open. 2023 Sep;7(5):823-840. doi: 10.1007/s41669-023-00419-w. Epub 2023 Jun 9. PMID 37296268
- [Derived] D'Haens G, Panaccione R, Baert F, Bossuyt P, Colombel JF, Danese S, Dubinsky M, Feagan BG, Hisamatsu T, Lim A, Lindsay JO, Loftus EV Jr, Panes J, Peyrin-Biroulet L, Ran Z, Rubin DT, Sandborn WJ, Schreiber S, Neimark E, Song A, Kligys K, Pang Y, Pivorunas V, Berg S, Duan WR, Huang B, Kalabic J, Liao X, Robinson A, Wallace K, Ferrante M. Risankizumab as induction therapy for Crohn's disease: results from the phase 3 ADVANCE and MOTIVATE induction trials. Lancet. 2022 May 28;399(10340):2015-2030. doi: 10.1016/S0140-6736(22)00467-6. PMID 35644154
- See also: Related info — https://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomized to receive 600mg risankizumab, 1200mg risankizumab or placebo during the double-blind, placebo-controlled Period 1. At Week 12, subjects who do not achieve clinical response were randomized into Period 2 to receive 180mg risankizumab, 360mg risankizumab or 1200mg risankizumab. Subjects who received placebo received 1200mg.
Pre-assignment Details: A total of 931 subjects were enrolled and included in the intent-to-treat (ITT) population; 850 of those had a baseline eligible Simple Endoscopic Score for Crohn's disease (SES-CD) of ≥ 6 (≥ 4 for isolated ileal disease) excluding the narrowing component and were included in the ITT1A population. This population was the primary population for both the United States (US) specific as well as the Global (Outside the US) efficacy analysis' of the 12-Week Induction Period.
Groups:
- Risankizumab 600mg (Induction Period 1): Participants randomized to receive risankizumab 600mg administered by intravenous (IV) infusion.
  risankizumab IV: Risankizumab administered by intravenous infusion
- Risankizumab 1200mg (Induction Period 1): Participants randomized to receive risankizumab 1200mg administered by intravenous (IV) infusion.
  risankizumab IV: Risankizumab administered by intravenous infusion
- Placebo (Induction Period 1): Participants randomized to receive placebo for risankizumab administered by intravenous (IV) infusion.
  placebo for risankizumab: Placebo for risankizumab administered by intravenous infusion
- Risankizumab 180mg (Induction Period 2): Participants with inadequate response at Week 12 in Period 1 randomized to receive risankizumab 180mg administered by subcutaneous (SC) injection in Period 2
- Risankizumab 360mg (Induction Period 2): Participants with inadequate response at Week 12 in Period 1 randomized to receive risankizumab 360mg administered by subcutaneous (SC) injection in Period 2.
  risankizumab SC: Risankizumab administered by subcutaneous (SC) injection
- Risankizumab 1200mg (Induction Period 2): Participants with inadequate response at Week 12 in Period 1 randomized to receive risankizumab 1200mg administered by intravenous infusion (IV) in Period 2.
  risankizumab IV: Risankizumab administered by intravenous infusion (IV)
- Placebo/Risankizumab IV (Induction Period 2): Participants who received placebo in Induction Period 1 received 1200 mg risankizumab by intravenous infusion (IV) at Weeks 12, 16, and 20.
  risankizumab IV: Risankizumab administered by intravenous infusion (IV)
Period: Period 1
Arm/Group | Risankizumab 600mg (Induction Period 1) | Risankizumab 1200mg (Induction Period 1) | Placebo (Induction Period 1) | Risankizumab 180mg (Induction Period 2) | Risankizumab 360mg (Induction Period 2) | Risankizumab 1200mg (Induction Period 2) | Placebo/Risankizumab IV (Induction Period 2)
Started (Randomized) | 373 | 372 | 186 | 0 | 0 | 0 | 0
Completed (Completed Period 1) | 365 | 366 | 163 | 0 | 0 | 0 | 0
Not Completed | 8 | 6 | 23 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Risankizumab 600mg (Induction Period 1) | Risankizumab 1200mg (Induction Period 1) | Placebo (Induction Period 1) | Risankizumab 180mg (Induction Period 2) | Risankizumab 360mg (Induction Period 2) | Risankizumab 1200mg (Induction Period 2) | Placebo/Risankizumab IV (Induction Period 2)
Started | 0 | 0 | 0 | 67 | 68 | 67 | 76
Completed (Completed study) | 0 | 0 | 0 | 62 | 65 | 64 | 74
Not Completed | 0 | 0 | 0 | 5 | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Consists of all subjects who received at least 1 dose of study medication.
Groups:
- Risankizumab 600mg (Period 1): Participants randomized to receive risankizumab 600mg administered by intravenous (IV) infusion.
  risankizumab IV: Risankizumab administered by intravenous infusion
- Risankizumab 1200mg (Period 1): Participants randomized to receive risankizumab 1200mg administered by intravenous (IV) infusion.
  risankizumab IV: Risankizumab administered by intravenous infusion
- Total: Total of all reporting groups
Arm/Group | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1) | Placebo (Period 1) | Total
Number analyzed (Participants) | 373 | 372 | 186 | 931
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 2 | 9
  Between 18 and 65 years | 355 | 350 | 175 | 880
  >=65 years | 15 | 18 | 9 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (13.22) | 37.6 (13.55) | 37.5 (13.51) | 37.9 (13.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 173 | 93 | 434
  Male | 205 | 199 | 93 | 497
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 18 | 10 | 41
  Not Hispanic or Latino | 360 | 354 | 176 | 890
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 68 | 75 | 32 | 175
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 10 | 13 | 9 | 32
  White | 291 | 279 | 144 | 714
  More than one race | 4 | 4 | 0 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: US Specific: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Clinical Remission
Description: The CDAI consists of 8 components; 7 are based on participant diary entries, participant interviews, physical examinations, measurement of body weight and height and 1 is based on laboratory analysis. CDAI clinical remission of Crohn's disease is defined as CDAI < 150.
Time Frame: Week 12
Population: Intent to Treat 1A Population: all randomized subjects who received at least one dose of study drug during the Induction Period 1, and had baseline eligible SES-CD of ≥ 6 (≥ 4 for isolated ileal disease) excluding the narrowing component.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 24.6 [18.2 to 31.0] | 45.2 [39.9 to 50.5] | 41.6 [36.3 to 46.8]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 20.7, 95% CI 2-sided [12.4 to 29.0]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 16.7, 95% CI 2-sided [8.5 to 24.9]

2. Primary Outcome: US Specific: Percentage of Participants With Endoscopic Response
Description: The SES-CD assesses endoscopic disease severity by evidence of active intestinal mucosal inflammation. Endoscopic response is defined as a decrease in SES-CD > 50% from Baseline (or for participants with isolated ileal disease and a Baseline SES-CD of 4, at least a 2-point reduction from Baseline).
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 12.0 [7.2 to 16.8] | 40.3 [35.0 to 45.6] | 32.1 [27.1 to 37.1]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 28.3, 95% CI 2-sided [21.2 to 35.4]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 20.3, 95% CI 2-sided [13.6 to 27.1]

3. Primary Outcome: Global Outside of US: Percentage of Participants With Clinical Remission
Description: Clinical remission is defined as using the average daily Stool Frequency (SF) ≤ 2.8 and not worse than Baseline AND average daily Abdominal Pain (AP) score ≤ 1 and not worse than Baseline.
Time Frame: Week 12
Population: Intent to Treat 1A Population: all randomized subjects who received at least one dose of study drug during the Induction Period 1 and had baseline eligible SES-CD of ≥ 6 (≥ 4 for isolated ileal disease) excluding the narrowing component.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 21.7 [15.6 to 27.8] | 43.5 [38.2 to 48.8] | 41.0 [35.8 to 46.2]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 21.9, 95% CI 2-sided [13.8 to 29.9]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 18.8, 95% CI 2-sided [10.8 to 26.8]

4. Primary Outcome: Global Outside of US: Percentage of Participants With Endoscopic Response
Description: as for outcome 2
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 12.0 [7.2 to 16.8] | 40.3 [35.0 to 45.6] | 32.1 [27.1 to 37.1]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 28.3, 95% CI 2-sided [21.2 to 35.4]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 20.3, 95% CI 2-sided [13.6 to 27.1]

5. Secondary Outcome: US Specific: Percentage of Participants With Clinical Remission
Description: as for outcome 3
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 21.7 [15.6 to 27.8] | 43.5 [38.2 to 48.8] | 41.0 [35.8 to 46.2]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 21.9, 95% CI 2-sided [13.8 to 29.9]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 18.8, 95% CI 2-sided [10.8 to 26.8]

6. Secondary Outcome: US Specific: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Clinical Response
Description: Crohn's Disease Activity Index (CDAI) is used to assess the symptoms of participants with Crohn's Disease. Higher CDAI scores indicate more severe disease. CDAI clinical response is defined as reduction of CDAI ≥ 100 points from baseline.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 25.2 [18.7 to 31.6] | 40.8 [35.5 to 46.0] | 37.2 [32.0 to 42.3]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 15.4, 95% CI 2-sided [7.2 to 23.7]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 11.2, 95% CI 2-sided [3.1 to 19.2]

7. Secondary Outcome: US Specific: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Clinical Response
Description: as for outcome 6
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 36.7 [29.6 to 43.9] | 59.7 [54.5 to 65.0] | 64.9 [59.8 to 70.0]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 23.1, 95% CI 2-sided [14.2 to 31.9]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 27.7, 95% CI 2-sided [19.0 to 36.4]

8. Secondary Outcome: US Specific: Change From Baseline of Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue
Description: The FACIT-Fatigue scale is a 13-item tool that measures an individual's level of fatigue during their usual daily activities over the past 7 days. Each of the fatigue and impact of fatigue items are measured on a four point Likert scale. The FACIT Fatigue Scale is the sum of the individual 13 scores and ranges from 0 to 52 where higher scores indicate better the quality of life. A positive change from baseline indicates improvement.
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 134 | 302 | 310
percentage of participants | 6.0 [4.4 to 7.7] | 11.2 [10.1 to 12.4] | 10.1 [9.0 to 11.3]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 5.2, 95% CI 2-sided [3.2 to 7.2]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 4.1, 95% CI 2-sided [2.1 to 6.1]

9. Secondary Outcome: US Specific: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Clinical Remission
Description: Crohn's Disease Activity Index (CDAI) is used to assess the symptoms of participants with Crohn's Disease. Higher CDAI scores indicate more severe disease. CDAI clinical remission of Crohn's disease is defined as CDAI < 150.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 10.3 [5.8 to 14.8] | 18.4 [14.3 to 22.6] | 18.9 [14.7 to 23.0]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p = 0.015, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 7.6, 95% CI 2-sided [1.5 to 13.7]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 8.4, 95% CI 2-sided [2.3 to 14.6]

10. Secondary Outcome: US Specific: Percentage of Participants With CDAI Clinical Response and Endoscopic Response
Description: Crohn's Disease Activity Index (CDAI) is used to assess the symptoms of participants with Crohn's Disease. Higher CDAI scores indicate more severe disease. CDAI clinical response is defined as reduction of CDAI ≥ 100 points from baseline.
  Endoscopic response was a decrease in Simplified Endoscopic Score for Crohn's Disease (SES-CD) > 50% from Baseline (or for subjects with isolated ileal disease and a Baseline SES-CD of 4, at least a 2 point reduction from Baseline).
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 5.7 [2.3 to 9.2] | 30.0 [25.1 to 34.9] | 23.0 [18.5 to 27.5]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 24.5, 95% CI 2-sided [18.5 to 30.5]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 17.3, 95% CI 2-sided [11.8 to 22.9]

11. Secondary Outcome: US Specific: Percentage of Participants With Stool Frequency (SF) Remission
Description: Stool Frequency (SF) remission is defined as an average daily SF <= 2.8 and not worse than baseline.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 29.8 [23.1 to 36.6] | 54.2 [48.8 to 59.5] | 54.0 [48.7 to 59.3]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 24.2, 95% CI 2-sided [15.7 to 32.7]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 23.6, 95% CI 2-sided [15.1 to 32.1]

12. Secondary Outcome: US Specific: Percentage of Participants With Abdominal Pain (AP) Remission
Description: The Abdominal Pain rating is an assessment that is graded from 0 to 3: 0= None, 1= Mild, 2= Moderate and 3= Severe. AP remission is defined as average daily AP score <= 1 and not worse than baseline.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 38.5 [31.2 to 45.7] | 59.6 [54.3 to 64.8] | 58.1 [52.9 to 63.4]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 21.2, 95% CI 2-sided [12.4 to 30.0]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 19.0, 95% CI 2-sided [10.1 to 27.8]

13. Secondary Outcome: US Specific: Percentage of Participants With Endoscopic Remission
Description: Endoscopic remission: SES-CD ≤ 4 and at least a 2 point reduction versus baseline and no subscore greater than 1 in any individual variable
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 9.1 [4.9 to 13.4] | 24.2 [19.6 to 28.7] | 23.9 [19.4 to 28.5]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 15.1, 95% CI 2-sided [9.0 to 21.2]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 15.4, 95% CI 2-sided [9.4 to 21.4]

14. Secondary Outcome: US Specific: Percentage of Participants With Enhanced Clinical Response
Description: Enhanced clinical response: ≥ 60% decrease in average daily SF and/or ≥ 35% decrease in average daily AP score and both not worse than Baseline, and/or clinical remission
Time Frame: Week 4
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 31.0 [24.1 to 37.9] | 46.0 [40.7 to 51.3] | 43.4 [38.1 to 48.6]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 14.9, 95% CI 2-sided [6.2 to 23.5]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 11.8, 95% CI 2-sided [3.2 to 20.3]

15. Secondary Outcome: US Specific: Percentage of Participants With Ulcer-Free Endoscopy
Description: Ulcer-free endoscopy: SES-CD ulcerated surface subscore of 0 in subjects with SES-CD ulcerated surface subscore ≥ 1 at Baseline
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 173 | 336 | 339
percentage of participants | 7.6 [3.6 to 11.5] | 21.0 [16.6 to 25.4] | 16.4 [12.4 to 20.3]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 13.7, 95% CI 2-sided [7.9 to 19.5]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 9.1, 95% CI 2-sided [3.7 to 14.5]

16. Secondary Outcome: US Specific: Percentage of Participants With Enhanced Clinical Response
Description: as for outcome 14
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 41.9 [34.6 to 49.3] | 62.8 [57.6 to 68.0] | 64.3 [59.2 to 69.4]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 21.0, 95% CI 2-sided [12.2 to 29.9]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 21.6, 95% CI 2-sided [12.8 to 30.4]

17. Secondary Outcome: US Specific: Percentage of Participants With Resolution of Extra-Intestinal Manifestations (EIMs), in Participants With EIMs at
Description: Manifestations of Crohn's disease in areas of the body other than the digestive tract, including eyes, skin, joints, mouth, and liver.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 64 | 140 | 158
percentage of participants | 20.5 [10.5 to 30.4] | 38.1 [30.0 to 46.1] | 43.7 [35.9 to 51.4]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p = 0.022, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 14.6, 95% CI 2-sided [2.1 to 27.0]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 23.7, 95% CI 2-sided [11.1 to 36.3]

18. Secondary Outcome: US Specific: Percentage of Participants With CD-Related Hospitalization
Description: Participants with at least one admission to the hospital due to Crohn's Disease.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 339 | 339
percentage of participants | 12.0 [7.2 to 16.8] | 3.3 [1.4 to 5.2] | 1.8 [0.4 to 3.2]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Chi-squared; Risk Difference (RD) = -8.7, 95% CI 2-sided [-13.9 to -3.5]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Chi-squared; Risk Difference (RD) = -10.2, 95% CI 2-sided [-15.2 to -5.2]

19. Secondary Outcome: US Specific: Percentage of Participants Without Draining Fistulas in Participants With Draining Fistulas at Baseline
Description: Participants without draining fistulas at Week 12 in participants who had draining fistulas at baseline.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 9 | 18 | 24
percentage of participants | 22.2 [0.0 to 49.4] | 27.8 [7.1 to 48.5] | 29.2 [11.0 to 47.4]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p = 1.00, Chi-squared; Risk Difference (RD) = 5.6, 95% CI 2-sided [-28.6 to 39.7]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p = 1.000, Chi-squared; Risk Difference (RD) = 6.9, 25% CI 2-sided [-25.7 to 39.6]

20. Secondary Outcome: Global Outside of US: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Clinical Remission
Description: The CDAI consists of 8 components; 6 are based on participant diary entries, participant interviews, and physical examinations, and 2 are based on laboratory analysis, and measurement of body weight and height. CDAI clinical remission of Crohn's disease is defined as CDAI < 150.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 24.6 [18.2 to 31.0] | 45.2 [39.9 to 50.5] | 41.6 [36.3 to 46.8]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 20.7, 95% CI 2-sided [12.4 to 29.0]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 16.7, 95% CI 2-sided [8.5 to 24.9]

21. Secondary Outcome: Global Outside of US: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Clinical Response
Description: as for outcome 6
Time Frame: Week 4
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 25.2 [18.7 to 31.6] | 40.8 [35.5 to 46.0] | 37.2 [32.0 to 42.3]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 15.4, 95% CI 2-sided [7.2 to 23.7]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 11.2, 95% CI 2-sided [3.1 to 19.2]

22. Secondary Outcome: Global Outside of US: Percentage of Participants With Clinical Remission
Description: as for outcome 3
Time Frame: Week 4
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 9.1 [4.9 to 13.4] | 21.0 [16.6 to 25.3] | 21.2 [16.9 to 25.6]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 11.5, 95% CI 2-sided [5.4 to 17.5]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 11.7, 95% CI 2-sided [5.7 to 17.8]

23. Secondary Outcome: Global Outside of US: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Clinical Response
Description: as for outcome 6
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 36.7 [29.6 to 43.9] | 59.7 [54.5 to 65.0] | 64.9 [59.8 to 70.0]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 23.1, 95% CI 2-sided [14.2 to 31.9]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 27.7, 95% CI 2-sided [19.0 to 36.4]

24. Secondary Outcome: Global Outside of US: Change From Baseline of Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue
Description: as for outcome 8
Time Frame: Week 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 134 | 302 | 310
units on a scale | 6.0 [4.4 to 7.7] | 11.2 [10.1 to 12.4] | 10.1 [9.0 to 11.3]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Mixed-Effect Model Repeat Measurement; LS Mean Difference = 5.2, 95% CI 2-sided [3.2 to 7.2]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Mixed-Effect Model Repeat Measurement; LS Mean Difference = 4.1, 95% CI 2-sided [2.1 to 6.1]

25. Secondary Outcome: Global Outside of US: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score
Description: The IBDQ is a 32-item (ranges 1 - 7) self-report questionnaire for patients with IBD to evaluate the patient reported outcomes across 4 dimensions: bowel symptoms (loose stools, abdominal pain), systemic symptoms (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability). The IBDQ total Score ranges from 32 to 224 with a higher score indicating better outcome.
Time Frame: Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 134 | 302 | 310
units on a scale | 23.6 [18.2 to 28.9] | 44.3 [40.6 to 48.0] | 43.0 [39.4 to 46.6]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Mixed-Effect Model Repeat Measurement; LS Mean Difference = 20.7, 95% CI 2-sided [14.3 to 27.1]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Mixed-Effect Model Repeat Measurement; LS Mean Difference = 19.4, 95% CI 2-sided [13.1 to 25.8]

26. Secondary Outcome: Global Outside of US: Percentage of Participants With Enhanced Clinical Response and Endoscopic Response
Description: Enhanced clinical response was defined as ≥ 60% decrease in average daily Stool Frequency and/or ≥ 35% decrease in average daily Abdominal Pain score and both not worse than baseline, and/or clinical remission. Endoscopic Response was defined as a decrease in Simplified Endoscopic Score for Crohn's Disease (SES-CD) > 50% from Baseline (or for subjects with isolated ileal disease and a Baseline SES-CD of 4, at least a 2 point reduction from Baseline).
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 8.0 [4.0 to 12.0] | 30.9 [25.9 to 35.8] | 23.2 [18.7 to 27.8]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 23.2, 95% CI 2-sided [16.8 to 29.6]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 15.2, 95% CI 2-sided [9.3 to 21.2]

27. Secondary Outcome: Global Outside of US: Percentage of Participants With Endoscopic Remission
Description: as for outcome 13
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 9.1 [4.9 to 13.4] | 24.2 [19.6 to 28.7] | 23.9 [19.4 to 28.5]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 15.1, 95% CI 2-sided [9.0 to 21.2]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 15.4, 95% CI 2-sided [9.4 to 21.4]

28. Secondary Outcome: Global Outside of US: Percentage of Participants With Enhanced Clinical Response
Description: as for outcome 14
Time Frame: Week 4
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 31.0 [24.1 to 37.9] | 46.0 [40.7 to 51.3] | 43.4 [38.1 to 48.6]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 14.9, 95% CI 2-sided [6.2 to 23.5]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 11.8, 95% CI 2-sided [3.2 to 20.3]

29. Secondary Outcome: Global Outside of US: Percentage of Participants With Ulcer-Free Endoscopy
Description: as for outcome 15
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 173 | 336 | 338
percentage of participants | 7.6 [3.6 to 11.5] | 21.0 [16.6 to 25.4] | 16.4 [12.4 to 20.3]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 13.7, 95% CI 2-sided [7.9 to 19.5]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 9.1, 95% CI 2-sided [3.7 to 14.5]

30. Secondary Outcome: Global Outside of US: Percentage of Participants With Enhanced Clinical Response
Description: as for outcome 14
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 41.9 [34.6 to 49.3] | 62.8 [57.6 to 68.0] | 64.3 [59.2 to 69.4]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 21.0, 95% CI 2-sided [12.2 to 29.9]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 21.6, 95% CI 2-sided [12.8 to 30.4]

31. Secondary Outcome: Global Outside of US: Percentage of Participants With Resolution of Extra-Intestinal Manifestations (EIMs), in Participants With EIMs at Baseline
Description: as for outcome 17
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 64 | 140 | 158
percentage of participants | 20.5 [10.5 to 30.4] | 38.1 [30.0 to 46.1] | 43.7 [35.9 to 51.4]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p = 0.022, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 14.6, 95% CI 2-sided [2.1 to 27.0]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted Risk Difference = 23.7, 95% CI 2-sided [11.1 to 36.3]

32. Secondary Outcome: Global Outside of US: Percentage of Participants With CD-Related Hospitalization
Description: Participants with at least one admission to the hospital due to Crohn's Disease.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 175 | 336 | 339
percentage of participants | 12.0 [7.2 to 16.8] | 3.3 [1.4 to 5.2] | 1.8 [0.4 to 3.2]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Mixed-Effect Model Repeat Measurement; LS Mean Difference = -8.7, 95% CI 2-sided [-13.9 to -3.5]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Mixed-Effect Model Repeat Measurement; LS Mean Difference = -10.2, 95% CI 2-sided [-15.2 to -5.2]

33. Secondary Outcome: Global Outside of US: Percentage of Participants Without Draining Fistulas in Participants With Draining Fistulas at Baseline
Description: Participants without draining fistulas at Week 12 in participants who had draining fistulas at baseline.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 9 | 18 | 24
percentage of participants | 22.2 [0.0 to 49.4] | 27.8 [7.1 to 48.5] | 29.2 [11.0 to 47.4]
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p = 1.000, Mixed-Effect Model Repeat Measurement; LS Mean Difference = 5.6, 95% CI 2-sided [-28.6 to 39.7]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p = 1.000, Mixed-Effect Model Repeat Measurement; LS Mean Difference = 6.9, 95% CI 2-sided [-25.7 to 39.6]

34. Secondary Outcome: Global Outside of US: Change From Baseline in Work Productivity and Impairment Questionnaire - Crohn's Disease (WPAI-CD) Overall Work Impairment
Description: WPAI: CD is a questionnaire used to evaluate lost productivity due to CD ; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Total work productivity impairment takes into account both hours missed due to CD symptoms and the patient's assessment of the degree to which CD affected their productivity while working (overall work impairment [OWI]). WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 65 | 156 | 162
units on a scale | -8.344 (3.5640) | -17.930 (2.3446) | -20.485 (2.3112)
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p = 0.024, Mixed-Effect Model Repeat Measurement; LS Mean Difference = -9.586, 95% CI 2-sided [-17.890 to -1.282]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p = 0.004, Mixed-Effect Model Repeat Measurement; LS Mean Difference = -12.141, 95% CI 2-sided [-20.390 to -3.892]

35. Secondary Outcome: Global Outside of US: Change From Baseline in Short Form-36 (SF-36) Physical Component Summary (PCS) Score
Description: The Short Form-36 Health Survey determined participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 comprise the physical component of the SF-36. Scores on each item were summed and averaged (range = 0-100); a positive change from Baseline indicates improvement.
Time Frame: Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Period 1) | Risankizumab 600mg (Period 1) | Risankizumab 1200mg (Period 1)
Number analyzed (Participants) | 134 | 302 | 309
units on a scale | 5.482 (0.5985) | 8.394 (0.4107) | 8.756 (0.4071)
Statistical Analysis 1: Comparison: Placebo (Period 1) vs Risankizumab 600mg (Period 1); Test type: Superiority; p < 0.001, Mixed-Effect Model Repeat Measurement; LS Mean Difference = 2.913, 95% CI 2-sided [1.512 to 4.313]
Statistical Analysis 2: Comparison: Placebo (Period 1) vs Risankizumab 1200mg (Period 1); Test type: Superiority; p < 0.001, Mixed-Effect Model Repeat Measurement; LS Mean Difference = 3.275, 95% CI 2-sided [1.877 to 4.672]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs (TEAEs) are from first dose of study drug until 140 days following last dose of study drug. The median duration of treatment for Period 1 with study drug for placebo and Risankizumab was 91.5 and 91 days respectively. For Period 2, the median duration of treatment with study drug for Risankizumab was 141 days.
Description: AEs/SAEs: As treated population: All randomized participants who took at least one does of study drug (Risankizumab/placebo), analyzed by the actual treatment the participant received.
Groups:
- Period 1 Placebo IV: Participants randomized to receive Placebo intravenous (IV) at Baseline, Weeks 4 and 8.
- Period 1 Risankizumab 600mg IV: Participants randomized to receive risankizumab 600mg intravenous (IV) at Baseline, Weeks 4 and 8.
- Period 1 Risankizumab 1200mg IV: Participants randomized to receive risankizumab 1200mg intravenous (IV) at Baseline, Weeks 4 and 8.
- Period 1 Risankizumab Total: Total Period 1 participants randomized into the Risankizumab treatment arm
- Period 2 Risankizumab 180mg SC: Participants randomized to receive risankizumab 180mg subcutaneously (SC) at Weeks 12 and 20.
- Period 2 Risankizumab 360mg SC: Participants randomized to receive risankizumab 360mg subcutaneously (SC) at Weeks 12 and 20.
- Period 2 Risankizumab 1200mg IV: Participants received risankizumab 1200mg intravenously at Weeks 12, 16, and 20.
- Period 2 Placebo/Risankizumab 1200mg IV: Participants who received placebo in Period 1 received 1200 mg risankizumab intravenously at Weeks 12, 16, and 20.
- Period 2 Risankizumab Total: Total Period 2 participants randomized into the Risankizumab treatment arm
Arm/Group | Period 1 Placebo IV | Period 1 Risankizumab 600mg IV | Period 1 Risankizumab 1200mg IV | Period 1 Risankizumab Total | Period 2 Risankizumab 180mg SC | Period 2 Risankizumab 360mg SC | Period 2 Risankizumab 1200mg IV | Period 2 Placebo/Risankizumab 1200mg IV | Period 2 Risankizumab Total
All-Cause Mortality (participants affected / at risk) | 2/186 | 0/373 | 0/372 | 0/745 | 0/67 | 0/68 | 0/67 | 0/76 | 0/278
Serious Adverse Events (participants affected / at risk) | 28/186 | 27/373 | 14/372 | 41/745 | 3/67 | 3/68 | 4/67 | 4/76 | 14/278
Other Adverse Events (participants affected / at risk) | 35/186 | 67/373 | 58/372 | 125/745 | 4/67 | 7/68 | 4/67 | 12/76 | 27/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1 Placebo IV (N=186) | Period 1 Risankizumab 600mg IV (N=373) | Period 1 Risankizumab 1200mg IV (N=372) | Period 1 Risankizumab Total (N=745) | Period 2 Risankizumab 180mg SC (N=67) | Period 2 Risankizumab 360mg SC (N=68) | Period 2 Risankizumab 1200mg IV (N=67) | Period 2 Placebo/Risankizumab 1200mg IV (N=76) | Period 2 Risankizumab Total (N=278)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINAL DISORDER (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 15 (16) | 5 (7) | 2 (2) | 7 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL NECROSIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ILEAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ILEAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
INTESTINAL STENOSIS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SUBILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TERMINAL ILEITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIVER DISORDER (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOOD ALLERGY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL WALL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABSCESS INTESTINAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
LEPTOSPIROSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VULVAL CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BODY TEMPERATURE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANKYLOSING SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FISTULA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENTAL DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OBSESSIVE-COMPULSIVE DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CALCULUS URINARY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1 Placebo IV (N=186) | Period 1 Risankizumab 600mg IV (N=373) | Period 1 Risankizumab 1200mg IV (N=372) | Period 1 Risankizumab Total (N=745) | Period 2 Risankizumab 180mg SC (N=67) | Period 2 Risankizumab 360mg SC (N=68) | Period 2 Risankizumab 1200mg IV (N=67) | Period 2 Placebo/Risankizumab 1200mg IV (N=76) | Period 2 Risankizumab Total (N=278)
ANAEMIA (Blood and lymphatic system disorders) | 5 (5) | 11 (11) | 9 (9) | 20 (20) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 7 (7)
CROHN'S DISEASE (Gastrointestinal disorders) | 10 (10) | 5 (5) | 4 (4) | 9 (9) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 10 (10) | 16 (17) | 13 (13) | 29 (30) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
NASOPHARYNGITIS (Infections and infestations) | 5 (5) | 22 (24) | 22 (24) | 44 (48) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 5 (5)
HEADACHE (Nervous system disorders) | 8 (8) | 24 (25) | 20 (27) | 44 (52) | 1 (2) | 3 (3) | 2 (3) | 5 (5) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT03105128/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT03105128/SAP_001.pdf